CLINICAL TRIAL: NCT06229860
Title: Impact of Personality on Adherence to Tyrosine Kinase Inhibitor Therapy in Patients with Chronic Myeloid Leukemia
Brief Title: Impact of Personality on Adherence to Tyrosine Kinase Inhibitor Therapy in Pts W/Chronic Myeloid Leukemia
Status: Recruiting | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Mahtab Jafari, Professor of Pharmaceutical Sciences & Equity Advisor, University of California, Irvine
Other Study IDs: 3709; UCI 23-110 (Other: UCI CFCCC)
Record Dates: First submitted 2024-01-17; First posted 2024-01-29 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Chronic Myeloid Leukemia; Chronic Phase Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult patients with CML in chronic phase (CML-CP)
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — In-person interview with the study coordinator to complete study questionnaire.

SUMMARY:
This is an observational pilot study to examine the association between a patient's personality and adherence to tyrosine kinase inhibitor therapy in patients with chronic myeloid leukemia.

DETAILED DESCRIPTION:
The purpose of this pilot study is to explore the association between personality and adherence to a specific type of oral cancer medication - tyrosine kinase inhibitor (TKI) - in patients with chronic myeloid leukemia (CML). 75 individuals with chronic phase CML who are being treated with TKIs will be recruited. Consenting patients will participate in a focused interview where TKI adherence, personality type, and quality of life and symptom burden will be assessed using validated questionnaires. Information on treatment response and the treating physician's perception of TKI adherence will be obtained from the electronic health record.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosed with chronic myeloid leukemia (CML) and in the chronic phase (CML-CP)
* Currently being treated with one of four cancer medications - imatinib, dasatinib, bosutinib, or nilotinib
* A patient at the UCI Chao Family Comprehensive Cancer Center (CFCCC), or
* A member of a patient support group organized by the CML Buster Foundation
* Do not meet any of the criteria listed under "Exclusion Requirements"

Exclusion Criteria:

* Unable to read and speak English
* Impaired decisional capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study populations include adult patients with CML in chronic phase (CML-CP) who are being treated with one of the four TKIs - imatinib, dasatinib, bosutinib, and nilotinib
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of adherence to TKI medication | Up to 1 year
  This will be measured by Morisky Medication Adherence Scale (MMAS), an 8-item tool related to adherence behavior include forgetfulness, stopping medication because of worsening of symptoms or improvement in health condition, and inconvenience of continuing medication. Each item is scored 0 or 1 depending on whether the patient answers yes or no, with a minimum score of 0 and maximum score of 8
Personality assessment | Up to 1 year
  Patient personality will be assessed using the Mini International Personality Item Pool (mini-IPIP) questionnaire. In the mini-IPIP, each of the five factors (openness, conscientiousness, extraversion, agreeableness and neuroticism) is assessed with four items, making a total of 20 items. Each item is scored on a scale of 1 through 5, with 1 indicating "very inaccurate" and 5 corresponding to "very accurate"
Assessment of quality of Life | Up to 1 year
  This will be measured by European Organisation of Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ C30). EORTC QLQ C30 includes 30 items that measure global health status, functioning, and symptoms.
Assessment of quality of Life and symptom burden | Up to 1 year
  This will be measured by European Organisation of Research and Treatment of Cancer Quality of Life Questionnaire Chronic Myeloid Leukemia -24 scales.(EROTC QLQ-CML 24). The EORTC QLQ CML 24 is a 24-item questionnaire developed exclusively to assess QoL issues in patients with CML

CONTACTS AND LOCATIONS:
Overall Officials: Mahtab Jafari, Pharm.D, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center University of California, Irvine, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No